CLINICAL TRIAL: NCT07132736
Title: Impact of Underwater Exercise Versus Regular Aerobic Exercise on Quality of Life and Power of Muscle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Kerolous Ishak Shehata, lecturer, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 11/6/2024-2025
Record Dates: First submitted 2025-06-25; First posted 2025-08-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Muscle Weakness | Patient; Quality of Life
Keywords: Under water exercise; Aerobic exercise; Muscle power; Quality of life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- underwater exercise (Experimental): Hydrotherapy uses the water as a supportive tool to reduce stress on muscles and joints during treatment.
  Performing exercises in warm water:
  * Relaxes muscles, improving range of motion.
  * Can significantly reduce chronic pain.
  * Supports weight, allowing for movements that may otherwise not be possible.
  Interventions: Device: Hubbard tank
- regular aerobic exercise (Experimental): Aerobic exercise is a physical activity that uses your body's large muscle groups, is rhythmic and repetitive. It increases your heart rate and how much oxygen your body uses. Examples of aerobic exercises include walking, cycling and swimming. It reduces your risk of heart disease, diabetes, high blood pressure and high cholesterol
  Interventions: Other: Mat on the ground

INTERVENTIONS:
Device: Hubbard tank — women will perform pelvic floor exercise and core stability exercise under water each session will be for 30 min
  Arms: underwater exercise
Other: Mat on the ground — women will perform core stability exercise and pelvic floor exercise on the mat for 30 min
  Arms: regular aerobic exercise

SUMMARY:
To investigate the Impact of underwater exercise versus regular aerobic exercise on quality of life and power of muscle

DETAILED DESCRIPTION:
To ensure statistical power and the reliability of results, the study will involve a sample size of sixty women between 16 and 50 years of age were randomly divided into an experimental and a study group (30 members each).

The experimental group will perform underwater exercise and the study group will perform regular aerobic exercise

ELIGIBILITY:
Inclusion Criteria:

1. BMI> 25
2. low muscle power
3. low quality of life
4. general fatigue

Exclusion Criteria:

1. BMI< 25
2. Polycystic ovarian syndrome
3. Chronic pelvic pain
4. Lumbar disc

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-28 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | The evaluation took place through study completion on 2 months
  A Visual Analogue Scale (VAS) is one of the pain rating scales and ranged from 0 point to 10 point. 0 point indicate that there is no pain, and 10 point indicates that their pain is maximum
Dynamomoter | The evaluation took place through study completion on 2 months
  A dynamometer is a device used to measure grip strength, providing a quantitative and objective assessment of muscular strength in the hand and forearm. percentage will be in newton, the higher of percentage indicate increase muscle power and lower of percentage indicate decrease muscle power
Psychological rating scale | The evaluation took place through study completion on 2 months
  Psychological rating scales are measurement instruments designed to assess and quantify various psychological constructs, such as attitudes, behaviors, and feelings. They allow researchers and clinicians to assign numerical values to abstract concepts, transforming subjective experiences into concrete data points

CONTACTS AND LOCATIONS:
Locations (1):
- Kerolous ishak shehata kelini, Amman, Jordan